CLINICAL TRIAL: NCT02660957
Title: Effectiveness of a Brief, Self-determination Intervention for Smoking Cessation (Immediate or Progressive) Among People Attending Emergency Departments: a Randomised Controlled Trial
Brief Title: Smoking Cessation Among People Attending A&E
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. LI William Ho Cheung, Associate Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: A&E
Record Dates: First submitted 2016-01-18; First posted 2016-01-21 (Estimated); Last update posted 2019-05-21 (Actual); Status verified 2019-05

CONDITIONS: Smoking
Keywords: Smoking cessation
MeSH Terms: conditions — Smoking; Smoking Cessation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- self-determination smoking cessation (Experimental): Subjects in the intervention group will be allowed to select their own schedules of quitting after discussing their situation with the counsellor (quit immediately (QI), or quit progressively (QP) with the ultimate goal of completing cessation over an acceptable period). Subjects in the intervention group will receive a self-help quitting leaflet published by the Hong Kong Council on Smoking and Health plus a series of brief interventions using the AWARD model.
  Interventions: Behavioral: self-determination smoking cessation
- health life (Placebo Comparator): Subjects in the placebo control group will receive a smoking cessation leaflet published by the Hong Kong Council on Smoking and Health (COSH), as will the intervention group. Moreover, subjects in the placebo control group will undergo a similar schedule of telephone follow-up as those in the intervention group. They will receive a 'placebo' intervention with a 'placebo booster' of the same duration on increasing physical activity and fruit and vegetable intake.
  Interventions: Other: placebo comparator

INTERVENTIONS:
Behavioral: self-determination smoking cessation — a self-help quitting leaflet plus a series of brief interventions using the AWARD model
  Arms: self-determination smoking cessation
Other: placebo comparator — suggest a healthy life style as a placebo comparator
  Arms: health life

SUMMARY:
The purpose of this study is to test the effectiveness of using a brief, self-determination intervention on smoking cessation (immediate or progressive) for people attending AEDs.

DETAILED DESCRIPTION:
Cigarette smoking, which causes serious damage to health resulting in many chronic problems including cancer, heart disease, stroke and lung disease, is the single most important, preventable cause of death and diseases. It is therefore crucial that healthcare professionals should promote smoking cessation and help patients quit. The Hong Kong government and community have put enormous efforts on raising tobacco tax, smoke-free legislation, law enforcement, health promotion campaigns and smoking cessation services. The prevalence of daily cigarette smokers has been decreasing from 23.3% in 1982 to 10.7 % in 2012, which is one of the lowest around the world. Nevertheless, about half of the smokers remain reluctant to even try giving up smoking.

Medical attention at Accident and Emergency Departments (AEDs) of smokers who are in physical discomfort can be developed as an excellent "teachable model" as it provides an invaluable opportunity to initiate smoking cessation. Smokers consulting doctors as an emergency are more liable to change their habits to improve their health. According to the Hospital Authority, about 2 million people attend AEDs in Hong Kong each year, of whom 68% are triaged as semi-urgent (level 4) and non-urgent (level 5). The average waiting time for a medical consultation varies among AEDs, but is generally longer than 30 min for triage level 4 and 1-2 h for level 5 - presenting healthcare professionals with a golden opportunity to advise smokers to quit and on the available smoking cessation programmes while they are waiting. However, most of the cessation programmes, including stage-matched interventions, generally take several to more than 30 minutes to implement and hence are not practicable or feasible in busy clinical settings. Indeed, the most common reason cited by healthcare professionals for being unable to help patients to quit smoking is the lack of time, because they are very busy and cannot spare even a few extra minutes to do so. Other barriers include a lack of training and experience, a lack of confidence in the effectiveness of the interventions, and the absence of incentives and deficiencies in support or requirements by hospital management that these programmes should be implemented. Moreover, our previous smoking cessation projects in outpatient clinics have revealed that many patients are too impatient to undergo a long intervention and some are reluctant to participate for fear that they might miss or experience delays in their medical consultation or other medical procedures. To address such problems, further studies are warranted to develop brief and effective interventions with simple, direct, strong, evidence-based warnings for patients who smoke.

Smoking is addictive and quitting is very difficult, with a high rate of relapse, particularly among those with high nicotine dependency. Our previous smoking cessation projects in outpatient clinics and the community have revealed that many smokers who are reluctant to quit are interested in reducing the number of cigarettes smoked per day. Therefore, another potential option would be to help smokers to reduce the number of cigarettes smoked gradually, with the ultimate goal of complete cessation. Several randomised controlled trials in the West have supported that smoking reduction interventions can help smokers first reduce and eventually quit smoking.

What investigators have achieved to date:

Investigators conducted a 'proof-of-principle' pilot randomised controlled trial on a very brief (<30 s) smoking cessation intervention with a 'one in two smokers will be killed by smoking' warning in medical outpatient clinics in Guangzhou. The results showed that more of the smokers who received this brief advice quit or reduced their smoking than did not. This pilot study suggested that even a very brief intervention on smoking cessation is better than no advice in the 'real world' practice for outpatient clinics. Moreover, the study demonstrated the feasibility and acceptability of the implementation of a very brief smoking cessation programme by healthcare professionals in busy clinical settings. In addition, the findings support the need for large randomised controlled trials of brief or minimal interventions with the 'one in two' warning.

In light of the above purpose, investigators designed a study with an experimental intervention for smoking cessation and a placebo comparator to act as control. Smokers randomly assigned to the intervention group were given a very brief (<30 s) smoking cessation intervention during telephone follow-ups with a 'one in two smokers will be killed by smoking' warning, and a self-help quitting leaflet published by the Hong Kong Council on Smoking and Health plus a series of brief interventions using the AWARD model. Whereas smokers randomly assigned to the placebo control group were given a 'placebo' intervention with a 'placebo booster' during telephone follow-ups (that had the same duration as the intervention), except that the content was about increasing physical activity and fruit and vegetable intake.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 years or above
* triaged as semi-urgent (level 4) or non-urgent (level 5)
* current smokers, either occasional or daily
* express a willingness to quit smoking

Exclusion Criteria:

* poor cognitive state or mental illness
* participation in other smoking cessation programmes or services

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1571 (Actual)
Dates: Start 2015-07; Primary Completion 2017-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
smoking quit rate change from baseline at 6-month follow-up between intervention and control group | 6-month follow-up
  The primary outcome is biochemically validated abstinence at 6 months.

SECONDARY OUTCOMES:
smoking quit rate change from baseline at 6-month and 12-month follow-up between intervention and control group | 6-month and 12-month follow-up
  self-reported 7-day point prevalence (pp) quit rate at 6 months and 12 months between the intervention and control group
smoking quit rate change from baseline at 12-month follow-up between intervention and control group | 12-month follow-up
  biochemically validated abstinence at 12 months.
smoking reduction rate change from baseline at 6-month and 12-month follow-up between intervention and control group | 6-month and 12-month follow-up
  self-reported reduction of ≥ 50% in cigarette consumption at 6 and 12 months between the intervention and control group
self-efficacy against tobacco change from baseline at 6-month and 12-month follow-up between intervention and control group | 6-month and 12-month follow-up
  self-efficacy against tobacco at 6 and 12 months follow-up between intervention and control group
quality of life change from baseline at 6-month and 12-month follow-up between intervention and control group | 6-month and 12-month follow-up
  quality of life at 6 and 12 months follow-up between intervention and control group

CONTACTS AND LOCATIONS:
Overall Officials: Ho Cheung William Li, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- Department of Accident and Emergency, United Christian Hospital, Hong Kong, China

REFERENCES:
- [Derived] Li WHC, Xia W, Wang MP, Cheung DYT, Cheung KY, Wong CKH, Lam TH. Effect of quitting immediately vs progressively on smoking cessation for smokers at emergency department in Hong Kong: A posteriori analysis of a randomized controlled trial. PLoS One. 2023 Jan 26;18(1):e0280925. doi: 10.1371/journal.pone.0280925. eCollection 2023. PMID 36701401
- [Derived] Li WHC, Ho KY, Wang MP, Cheung DYT, Lam KKW, Xia W, Cheung KY, Wong CKH, Chan SSC, Lam TH. Effectiveness of a Brief Self-determination Theory-Based Smoking Cessation Intervention for Smokers at Emergency Departments in Hong Kong: A Randomized Clinical Trial. JAMA Intern Med. 2020 Feb 1;180(2):206-214. doi: 10.1001/jamainternmed.2019.5176. PMID 31790546